CLINICAL TRIAL: NCT05096091
Title: International Study on COVID-19 Vaccine to Assess Immunogenicity, Reactogenicity and Efficacy (InVITE)
Acronym: InVITE
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Partnership for Clinical Research in Guinea/Partenariat de Recherche Clinique en Guinée (PREGUI) (Unknown); Partnership for Research on Ebola Virus in Liberia (PREVAIL) (Network); University Clinical Research Center, Mali (Other); Onom Foundation and Liver Center (Unknown); Mexican Emerging Infectious Diseases Clinical Research Network (Network); Ina-Respond (Other)
Responsible Party: Sponsor
Other Study IDs: InVITE 01
Record Dates: First submitted 2021-10-26; First posted 2021-10-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, and nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
InVITE is funded by NIAID and is conducted in multiple international sites (approximately 20 sites across 7 countries).

This is a study of adults who receive locally available COVID-19 vaccines through local vaccination programs. Persons will be enrolled within one day (before or after) of receipt of a COVID-19 vaccine. The study will enroll participants who receive COVID-19 vaccination at local clinics and/or study sites.

DETAILED DESCRIPTION:
This is a multicenter study of COVID-19 vaccine immunogenicity and durability, and breakthrough serious acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infections in people who receive a COVID-19 vaccine through their country's national vaccination programs. Participants will be enrolled upon signing the informed consent within a day of receipt of a COVID-19 vaccine (before or after). The study team will not be administering the vaccine; receipt of vaccine will be provided through each country's vaccine program. Blood specimens will be collected to measure the immune response to the vaccine. Participants may be asked to contact study staff at any time during the study for evaluation if they develop symptoms consistent with SARS-CoV-2 infection, at which time they will be counseled about the need for a medical evaluation that may include collection of an upper airway swab for diagnosis (and research) and a blood sample for research. Infections will be confirmed by molecular or antigen (Ag) testing at the time of symptoms, and swabs will be collected and stored for viral sequencing and analyses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Ability to provide informed consent.
* Enrollment within one day (before or after) of receipt of COVID-19 vaccine.
* Willingness to be evaluated (including collection of blood and nasopharyngeal samples) during the prescribed study visits and/or during acute illness consistent with SARS-CoV-2 infection during the study period.
* Willingness to allow storage of biological samples for research testing as outlined in this protocol.

Exclusion Criteria:

* Any acute or chronic condition that, in the opinion of the investigator, is a contraindication to participation in this study; for example, acute febrile illness.
* Inability to comply with study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be people who are about to receive or have already received a Coronavirus disease 2019 (COVID-19) vaccine through the local vaccination program.
Sampling Method: Probability Sample
Enrollment: 5399 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
1. To characterize immunogenicity (by measurement of anti-Spike [S] antibody [Ab]) of available COVID-19 vaccines in the overall study population, in each of the countries and in defined subgroups | 2 months
  Measured by amount of Anti-S Ab at 2 months after completion of vaccine regimen.

SECONDARY OUTCOMES:
Evaluate duration of immunogenicity | 1 day, 2 months, 10 months
  Measured by Anti-S Ab at different specific timepoints
Evaluate immunogenicity in predefined subgroups (by age, body mass index [BMI], comorbidities, HIV, breakthrough infection, or evidence of prior infection with SARS-CoV-2). | 1 day, 2 months, 10 months
  Measured by levels of Anti-S Ab in predefined subgroups.
Characterize virus causing breakthrough infections using viral genomic sequencing. | 1 day
  Measured from sequencing to characterize SARS-CoV-2 variants
Compare immunogenicity between different vaccines. | 2 months
  Measured by Anti-S Ab levels at 2 months post-vaccine regimen
Evaluate infection rates after vaccination. | 1 day
  Measured by levels of anti-nucleocapsid Ab

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ridzon, MD, Study Director — National Institute of Allergy and Infectious Diseases (NIAID); Irini Sereti, MD, Study Director — National Institute of Allergy and Infectious Diseases (NIAID); Sally Hunsberger, PhD, Study Director — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (11):
- National Institute for Biomedical Research/Institut National de Recherche Biomédicale (INRB), Gombe, Kinshasa City, Democratic Republic of the Congo
- Partnership for Clinical Research in Guinea/Partenariat de Recherche Clinique en Guinée (PREGUI), Conakry, Guinea
- National Institute of Health Research and Development (NIHRD), Ministry of Health, Republic of Jakarta - RSU Kabupaten Tangerang, Tangerang, Indonesia
- Partnership for Research in Vaccines and Infectious Diseases in Liberia (PREVAIL) - Duport Road Health Center, Monrovia, Liberia
- University Clinical Research Center (UCRC) University of Sciences, Techniques and Technologies of Bamako, Bamako, Mali
- Mexico (5):
  - Hospital Regional de Alta Especialidad "Ciudad Salud" HRAE-CS, Tapachula, Chiapas
  - Hospital General Dr. Manuel Gea Gonzalez (HGMGG), Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (INCMNSZ),, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias (INER), Mexico City
  - Hospital General Dr. Aurelio Valdivieso (HGAV), Oaxaca City
- Onom Foundation and Liver Center, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laverdure S, Kazadi D, Kone K, Callier V, Dabitao D, Dennis D, Haidara MC, Hunsberger S, Mbaya OT, Ridzon R, Sereti I, Shaw-Saliba K; InVITE Study Team. SARS-CoV-2 seroprevalence in vaccine-naive participants from the Democratic Republic of Congo, Guinea, Liberia, and Mali. Int J Infect Dis. 2024 May;142:106985. doi: 10.1016/j.ijid.2024.106985. Epub 2024 Feb 28. PMID 38417612
- See also: SARS-CoV-2 seroprevalence in vaccine-naïve participants from the Democratic Republic of Congo, Guinea, Liberia, and Mali — https://pubmed.ncbi.nlm.nih.gov/38417612/